CLINICAL TRIAL: NCT00082888
Title: Phase II Evaluation of FTI (R115777) in Treatment of Relapsed and Refractory Lymphoma
Brief Title: Tipifarnib in Treating Patients With Relapsed or Refractory Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02849; NCI-2012-02849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LS038B; LS038B (Other: Mayo Clinic); 6246 (Other: CTEP); P30CA015083 (NIH); P50CA097274 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Results first posted 2011-12-07 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Anaplastic Large Cell Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Nodal Marginal Zone Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult T-Cell Leukemia/Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tipifarnib

ARMS (1):
- Treatment (tipifarnib) (Experimental): Patients receive tipifarnib PO BID on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Tipifarnib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Tipifarnib — Given PO
  Other Names: R115777; Zarnestra

SUMMARY:
This phase II trial studies how well tipifarnib works in treating patients with relapsed or refractory non-Hodgkin's lymphoma. Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Tipifarnib may be an effective treatment for non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess tumor response to R115777 (tipifarnib) in patients with relapsed aggressive non-Hodgkin's lymphoma. (Permanently closed to accrual 6/28/06) II. To assess tumor response to R115777 in patients with relapsed indolent non-Hodgkin's lymphoma. (Permanently closed to accrual 9/26/07) III. To assess tumor response to R115777 in patients with uncommon non-Hodgkin's lymphomas.

IV. To evaluate toxicity associated with this regimen in patients with relapsed non-Hodgkin's lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate known and unknown molecular markers that may predict for response to R115777 in lymphoma tissue.

OUTLINE:

Patients receive tipifarnib orally (PO) twice daily (BID) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven relapsed or refractory lymphomas; previous biopsies =< 6 months prior to treatment on this protocol will be acceptable as long as there has not been intervening therapy; if the patient has received therapy for non-Hodgkin's disease (NHL) between the time of the last biopsy and this protocol, then a re-biopsy is necessary
* STUDY 1: Aggressive lymphomas (permanently closed to accrual 6/28/06):

  * Transformed lymphomas
  * Diffuse large B cell lymphoma
  * Mantle cell lymphoma
  * Follicular lymphoma grade III STUDY 2: Indolent lymphomas (permanently closed to accrual 9/26/07)
  * Small lymphocytic lymphoma/chronic lymphocytic leukemia
  * Follicular lymphoma, grades 1, 2
  * Extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue (MALT) type
  * Nodal marginal zone B-cell lymphoma
  * Splenic marginal zone B-cell lymphoma

STUDY 3: Uncommon lymphomas:

* Peripheral T cell lymphoma, unspecified
* Anaplastic large cell lymphoma (T and null cell type)
* Lymphoplasmacytic lymphoma
* Mycosis fungoides/ Sezary syndrome
* Relapsed Hodgkin's disease (patients must be previously treated and either have had a transplant or not be eligible for a transplant)

  * Previously treated (no limitations on the number of prior therapies); patients with aggressive lymphoma (Study 1 - permanently closed to accrual 6/28/06) should have received or be ineligible for potentially curable therapy including stem cell transplant
  * MEASURABLE DISEASE: Must have at least one lesion that has a single diameter of >= 2 cm or tumor cells in the blood >= 5 x10^9/L
  * Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
  * Absolute neutrophil count >=1000/mm^3
  * Platelet count >= 75,000
  * Hemoglobin >= 9 g/dL
  * Total bilirubin =< 2 x upper limit of normal (ULN) (if > 2 x ULN direct bilirubin is required and should be =< 1.5 x ULN)
  * Aspartate aminotransferase (AST) =< 3 x ULN (=< 5 x ULN if liver involvement is present)
  * Serum creatinine =< 2 x ULN
  * Expected survival >= 3 months
  * Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent
  * Capable of swallowing intact study medication tablets
  * Capable of following directions regarding taking study medication, or has a daily caregiver who will be responsible for administering study medication

Exclusion Criteria:

* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
  * NOTE: The effects of R115777 on the developing human fetus at the recommended therapeutic dose are unknown
* Life-threatening illness (unrelated to tumor)
* Ongoing radiation therapy or radiation therapy =< 3 weeks prior to study registration unless the acute side effects associated with such therapy are resolved
* Therapy with myelosuppressive chemotherapy, cytotoxic chemotherapy, or biologic therapy =< 3 weeks (6 weeks for nitrosourea or mitomycin C) or corticosteroids =< 2 weeks, prior to starting R11577; patients may be on corticosteroids or tapering off them up until the day they start R11577 as long as it is clear that they are not having a tumor response to the steroids or that the steroids would confuse the interpretation of response to R11577; patients may be receiving stable (not increased within the last month) chronic doses of corticosteroids with a maximum dose of 20 mg of prednisone per day if they are being given for disorders other than lymphoma such as rheumatoid arthritis, polymyalgia rheumatica, adrenal insufficiency, or intractable symptoms of lymphoma
* Peripheral neuropathy >= grade 3
* Serious non-malignant disease such as active infection or other condition which in the opinion of the investigator would compromise other protocol objectives
* Presence of central nervous system (CNS) lymphoma
* Other active malignancies
* Once a patient begins FTI (tipifarnib) treatment, the addition of other cancer treatment will confound the assessment of efficacy and therefore is not allowed; this restriction precludes the addition of cytotoxic, immunologic agents, radiotherapy, or an increase in corticosteroid dose while the patient is in the treatment phase of this protocol
* Known to be human immunodeficiency virus (HIV) positive; HIV testing is not required but should be done if clinically indicated; HIV patients are excluded because of concerns regarding excess risk of complications of immunosuppressive therapy regimens
* Known allergy to imidazole drugs such as clotrimazole, ketoconazole, miconazole, econazole, fenticonazole, sulconazole, tioconazole, or terconazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2004-03-24 (Actual); Primary Completion 2009-05-20 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Witzig, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Witzig TE, Tang H, Micallef IN, Ansell SM, Link BK, Inwards DJ, Porrata LF, Johnston PB, Colgan JP, Markovic SN, Nowakowski GS, Thompson CA, Allmer C, Maurer MJ, Gupta M, Weiner G, Hohl R, Kurtin PJ, Ding H, Loegering D, Schneider P, Peterson K, Habermann TM, Kaufmann SH. Multi-institutional phase 2 study of the farnesyltransferase inhibitor tipifarnib (R115777) in patients with relapsed and refractory lymphomas. Blood. 2011 Nov 3;118(18):4882-9. doi: 10.1182/blood-2011-02-334904. Epub 2011 Jul 1. PMID 21725056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 medical clinics in the United States between March 2004 to November 2008.
Groups:
- Aggressive B-cell NHL Group: Patients with aggressive B-cell NHL receive 300mg twice a day for 21 days. Cycle length is 28 days. After cycle 1, may increase the dose to 400mg twice a day or 600mg twice a day at physician discretion.
- Indolent B-cell NHL Group: Patients with indolent B-cell NHL receive 300mg twice a day for 21 days. Cycle length is 28 days. After cycle 1, may increase the dose to 400mg twice a day or 600mg twice a day at physician discretion.
- HL/T-cell Lymphoma Group: Patients with HL/T-cell lymphoma receive 300mg twice a day for 21 days. Cycle length is 28 days. After cycle 1, may increase the dose to 400mg twice a day or 600mg twice a day at physician discretion.
Period: Overall Study
Arm/Group | Aggressive B-cell NHL Group | Indolent B-cell NHL Group | HL/T-cell Lymphoma Group
Started | 42 | 15 | 36
Completed | 41 | 15 | 36
Not Completed | 1 | 0 | 0
Not completed — Ineligible | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants are included in this baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aggressive B-cell NHL Group | Indolent B-cell NHL Group | HL/T-cell Lymphoma Group | Total
Number analyzed (Participants) | 42 | 15 | 36 | 93
Age, Continuous [Median (Full Range); unit: years] | 66.5 [44.0 to 91.0] | 64.0 [45.0 to 83.0] | 48.5 [18.0 to 91.0] | 62 [18 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 14 | 42
  Male | 24 | 5 | 22 | 51

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Confirmed Response (Complete Response, Unconfirmed Complete Response, or Partial Response) During the First 6 Courses of Treatment
Description: Confirmed response is at least a 50% decrease in the sum of the products of the greatest diameters (SPD) of the six largest dominant nodes or nodal masses and no increase in the size of other nodes, liver, or spleen and splenic and hepatic nodules must regress by at least 50% in the SPD and no new sites of disease.
Time Frame: During the first 6 cycles of treatment
Population: All participants are included in this analysis.
Measure: Number; unit: Proportion of participants
Arm/Group | Aggressive B-cell NHL Group | Indolent B-cell NHL Group | HL/T-cell Lymphoma Group
Number analyzed (Participants) | 42 | 15 | 36
Proportion of participants | 0.17 | 0.07 | 0.31

2. Secondary Outcome: Overall Survival
Description: Overall survival time was defined as the time from registration to the date of death or last follow-up.
Time Frame: Up to 2 years
Population: All participants are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aggressive B-cell NHL Group | Indolent B-cell NHL Group | HL/T-cell Lymphoma Group
Number analyzed (Participants) | 42 | 15 | 36
months | 6.4 [4.1 to 10.7] | 20.6 [16.6 to NA] — The 95% confidence interval upper limit was not reached (i.e., insufficient number of participants with events). | 19.7 [9 to 60]

3. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the number of months from registration to the date of disease progression with patients being progression-free being censored on the date of their last evaluation. Progression is defined as ≥50 % increase from nadir in the SPD of any previously identified abnormal node for partial responders or nonresponders or appearance of any new lesion during or at the end of therapy.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aggressive B-cell NHL Group | Indolent B-cell NHL Group | HL/T-cell Lymphoma Group
Number analyzed (Participants) | 42 | 15 | 36
months | 2.8 [1.7 to 4.2] | 5.2 [4 to 9.2] | 3.2 [1.9 to 5.8]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients that have achieved an objective response as the date at which the patient's objective status is first noted to be either a complete response (CR) or partial response (PR) to the date progression (PD) is documented. CR:Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy PR:≥50% decrease in SPD of the six largest dominant nodes or nodal masses. PD:≥50 % increase from nadir in the SPD of any previously identified abnormal node for PRs or nonresponders or appearance of any new lesion during or at the end of therapy.
Time Frame: up to 2 years
Population: Patients who had a response were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aggressive B-cell NHL Group | Indolent B-cell NHL Group | HL/T-cell Lymphoma Group
Number analyzed (Participants) | 7 | 1 | 11
months | 11.3 [4.9 to 17.1] | 2 | 7.5 [3.2 to 29.8]

5. Secondary Outcome: Number of Patients Who Experienced Grade 3 or 4 Toxicities
Description: Number of patients that experienced a grade 3 or 4 toxicity (adverse events considered at least possibly related to Tipifarnib) as measured by NCI (National Cancer Institute) CTCAE (Common Terminology Criteria for Adverse Events) v3.0.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL(Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.).
  Grade 4: Life-threatening consequences; urgent intervention indicated.
Time Frame: Up to 56 days
Population: Only eligible participants are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Aggressive B-cell NHL Group | Indolent B-cell NHL Group | HL/T-cell Lymphoma Group
Number analyzed (Participants) | 41 | 15 | 36
Participants | 32 | 8 | 24

ADVERSE EVENTS:
Description: Only eligible participants are included in this analysis.
Arm/Group | Aggressive B-cell NHL Group | Indolent B-cell NHL Group | HL/T-cell Lymphoma Group
All-Cause Mortality (participants affected / at risk) | 34/41 | 9/15 | 27/36
Serious Adverse Events (participants affected / at risk) | 27/41 | 4/15 | 20/36
Other Adverse Events (participants affected / at risk) | 38/41 | 15/15 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggressive B-cell NHL Group (N=41) | Indolent B-cell NHL Group (N=15) | HL/T-cell Lymphoma Group (N=36)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (7) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder infection(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colitis, infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Sepsis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Soft tissue infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Wound infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 8 (8) | 2 (3) | 7 (8)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 15 (17) | 3 (4) | 9 (12)
Platelet count decreased (Investigations) | 8 (8) | 4 (5) | 8 (11)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (5)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggressive B-cell NHL Group (N=41) | Indolent B-cell NHL Group (N=15) | HL/T-cell Lymphoma Group (N=36)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 32 (121) | 14 (43) | 26 (136)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Flashing vision (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 11 (16) | 5 (14) | 12 (20)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 1 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (7)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 6 (16) | 12 (18)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (5) | 2 (3)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (5)
Edema limbs (General disorders) | 5 (6) | 1 (1) | 0 (0)
Fatigue (General disorders) | 32 (92) | 14 (51) | 32 (188)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (4)
General symptom (General disorders) | 0 (0) | 0 (0) | 1 (2)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (5) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 2 (5) | 1 (1)
Catheter related infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection - Neck(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Mucosal infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pleural infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Sinusitis(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection(unknown ANC) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 8 (31) | 1 (6) | 11 (23)
Aspartate aminotransferase increased (Investigations) | 14 (49) | 4 (9) | 8 (18)
Blood bilirubin increased (Investigations) | 5 (5) | 4 (10) | 5 (7)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 12 (58) | 5 (16) | 5 (55)
Leukocyte count decreased (Investigations) | 21 (64) | 7 (24) | 15 (36)
Lymphocyte count decreased (Investigations) | 2 (4) | 1 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 17 (42) | 8 (20) | 15 (49)
Platelet count decreased (Investigations) | 29 (123) | 8 (43) | 23 (137)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 2 (4) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 2 (6) | 3 (3)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 7 (7) | 2 (2) | 4 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 3 (4)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (5) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 4 (8) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 3 (4) | 2 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (72) | 6 (12) | 11 (134)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (6) | 1 (1)
Confusion (Psychiatric disorders) | 4 (4) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 3 (6) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (2) | 2 (2)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (13)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 10 (22) | 2 (4) | 13 (55)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (12)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less